CLINICAL TRIAL: NCT03346070
Title: A Phase 4 Randomized, Active-Comparator Controlled Trial to Study the Efficacy and Safety of Sugammadex (MK-8616) for the Reversal of Neuromuscular Blockade Induced by Either Rocuronium Bromide or Vecuronium Bromide in Morbidly Obese Subjects
Brief Title: Efficacy and Safety of Sugammadex Dosed According to Actual Body Weight (ABW) or Ideal Body Weight (IBW) in Reversal of Neuromuscular Blockade (NMB) in Morbidly Obese Participants (MK-8616-146)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 8616-146; 2017-000188-33 (EudraCT Number); MK-8616-146 (Other: Merck Protocol Number)
Record Dates: First submitted 2017-11-15; First posted 2017-11-17 (Actual); Results first posted 2019-12-23 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Neuromuscular Blockade
MeSH Terms: interventions — Sugammadex; Neostigmine; Glycopyrrolate; Rocuronium; Vecuronium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Sugammadex 2 mg/kg ABW (Experimental): Following administration of NMBA, participants received a single intravenous (i.v.) bolus of Sugammadex at 2 mg/kg as determined utilizing participant ABW. A treatment dose of 2 mg/kg was used for reversal of moderate NMB.
  Interventions: Drug: Sugammadex 2 mg/kg ABW; Drug: Rocuronium or Vecuronium
- Sugammadex 2 mg/kg IBW (Experimental): Following administration of NMBA, participants received a single i.v. bolus of Sugammadex at 2 mg/kg as determined utilizing participant IBW. A treatment dose of 2 mg/kg was used for reversal of moderate NMB.
  Interventions: Drug: Sugammadex 2 mg/kg IBW; Drug: Rocuronium or Vecuronium
- Sugammadex 4 mg/kg ABW (Experimental): Following administration of NMBA, participants received a single i.v. bolus of Sugammadex at 4 mg/kg as determined utilizing participant ABW. A treatment dose of 4 mg/kg was used for reversal of deep NMB.
  Interventions: Drug: Sugammadex 4 mg/kg ABW; Drug: Rocuronium or Vecuronium
- Sugammadex 4 mg/kg IBW (Experimental): Following administration of NMBA, participants received a single i.v. bolus of Sugammadex at 4 mg/kg as determined utilizing participant IBW. A treatment dose of 4 mg/kg was used for reversal of deep NMB.
  Interventions: Drug: Sugammadex 4 mg/kg IBW; Drug: Rocuronium or Vecuronium
- Neostigmine/Glycopyrrolate (Active Comparator): Following administration of NMBA, participants received a single i.v. bolus containing both Neostigmine (50 µg/kg; up to 5 mg maximum dose) and Glycopyrrolate (10 µg/kg; up to 1 mg maximum dose) as determined utilizing participant ABW. Neostigmine/Glycopyrrolate was used for reversal of moderate NMB. Active comparator treatment for reversal for deep NMB was not available.
  Interventions: Drug: Neostigmine + Glycopyrrolate; Drug: Rocuronium or Vecuronium

INTERVENTIONS:
Drug: Sugammadex 2 mg/kg ABW — Following administration of NMBA (Rocuronium or Vecuronium) to achieve moderate NMB, participants received a single i.v. bolus of Sugammadex (2 mg/kg by ABW) for reversal of moderate NMB.
  Moderate NMB is defined as the reappearance of a second twitch (T2) in response to TOF stimulations.
  Other Names: MK-8616
  Arms: Sugammadex 2 mg/kg ABW
Drug: Sugammadex 2 mg/kg IBW — Following administration of NMBA (Rocuronium or Vecuronium) to achieve moderate NMB, participants received a single i.v. bolus of Sugammadex (2 mg/kg by IBW) for reversal of moderate NMB.
  Moderate NMB is defined as the reappearance of T2 in response to TOF stimulations.
  Other Names: MK-8616
  Arms: Sugammadex 2 mg/kg IBW
Drug: Sugammadex 4 mg/kg ABW — Following administration of NMBA (Rocuronium or Vecuronium) to achieve deep NMB, participants received a single i.v. bolus of Sugammadex (4 mg/kg by ABW) for reversal of deep NMB.
  Deep NMB is defined as no response to TOF stimulations (TOF=0) and a detection target of 1-2 post-tetanic counts (PTCs).
  Other Names: MK-8616
  Arms: Sugammadex 4 mg/kg ABW
Drug: Sugammadex 4 mg/kg IBW — Following administration of NMBA (Rocuronium or Vecuronium) to achieve deep NMB, participants will receive a single i.v. bolus of Sugammadex (4 mg/kg by IBW) for reversal of deep NMB.
  Deep NMB is defined as no response to TOF stimulations (TOF=0) and a detection target of 1-2 post-tetanic counts (PTCs).
  Other Names: MK-8616
  Arms: Sugammadex 4 mg/kg IBW
Drug: Neostigmine + Glycopyrrolate — Following administration of NMBA (Rocuronium or Vecuronium) to achieve moderate NMB, participants received a single i.v. bolus of Neostigmine (50 µg/kg; 5 mg maximum) and Glycopyrrolate (10 µg/kg; 1 mg maximum), dosed according to participant ABW for reversal of moderate NMB.
  Moderate NMB is defined as the reappearance of T2 in response to TOF stimulations.
  Arms: Neostigmine/Glycopyrrolate
Drug: Rocuronium or Vecuronium — To achieve NMB, participants received steroidal NMBA Rocuronium Bromide or Vecuronium Bromide administered via i.v. infusion and dosed according to participant ABW. NMBAs were concomitant medications used per label as adjunct to general anesthesia.

SUMMARY:
The purpose of this trial is to evaluate the safety and efficacy of Sugammadex when administered according to actual body weight (ABW) as compared to ideal body weight (IBW) for the reversal of both moderate and deep neuromuscular blockade (NMB) induced by either Rocuronium or Vecuronium in morbidly obese participants. The primary hypothesis of this investigation is that, compared to obese participants dosed based on IBW, obese participants receiving Sugammadex according to ABW will demonstrate a faster time to recovery to a Train Of Four (TOF) ratio of ≥0.9 (i.e. faster NMB reversal), pooled across NMB depth and type of neuromuscular blocking agent (NMBA; Rocuronium or Vecuronium) administered.

ELIGIBILITY:
Inclusion Criteria:

* Have BMI ≥40 kg/m² (morbidly obese).
* Be categorized as American Society of Anesthesiologists (ASA) Physical Status Class 3
* Have a planned surgical procedure that requires neuromuscular block with either rocuronium or vecuronium.
* Have a planned surgical procedure (e.g., gastrointestinal, urologic, or laparoscopic procedures) that in the opinion of the investigator does not preclude maintenance of moderate or deep depth of NMB throughout the case (maintained by re-dosing or continuous infusion).
* Have a planned surgical procedure that would allow objective neuromuscular monitoring techniques to be applied with access to the arm for neuromuscular transmission monitoring.
* If female, who is not of reproductive potential, be one of the following: 1) postmenopausal (defined as at least 12 months with no menses in women ≥45 years of age; 2) has had a hysterectomy and/or bilateral oophorectomy, bilateral salpingectomy, or bilateral tubal ligation/occlusion at least 6 weeks prior to screening; 3) has a congenital or acquired condition that prevents childbearing; or 4) is undergoing surgical sterilization as the planned surgical procedure associated with participation in this study (e.g., hysterectomy or tubal ligation).
* If female, who is sexually active and of child-bearing potential, agrees to use a medically accepted method of contraception through seven days after receiving protocol-specified medication. Please note the following: 1) Medically accepted methods of contraception include condoms (male or female) with a spermicidal agent, diaphragm or cervical cap with spermicide, medically prescribed intrauterine device (IUD), inert or copper-containing IUD, surgical sterilization (e.g., hysterectomy or tubal ligation); 2) Abstinence (relative to heterosexual activity) can be used as the sole method of contraception if it is consistently employed as the subject's preferred and usual lifestyle and if considered acceptable by local regulatory agencies and Human Subjects Protection Review Boards; 3 Periodic abstinence (e.g., calendar, ovulation, sympto-thermal, post-ovulation methods, etc.) and withdrawal are not acceptable methods of contraception; 4) If a contraceptive method listed above is restricted by local regulations/guidelines, then it does not qualify as an acceptable method of contraception for subjects participating at sites in this country/region.
* Be able to provide (or the subject's legally authorized representative in accordance with local requirements), written informed consent for the trial. The participant or legally authorized representative may also provide consent for Future Biomedical Research.

Exclusion Criteria:

* Have an actual body weight <100 kg.
* Have a pacemaker or automatic implantable cardioverter-defibrillator that precludes the assessment of bradycardia or arrhythmias.
* Have a medical condition or surgical procedure that precludes reversal of neuromuscular block at the end of surgery.
* Have neuromuscular disorder(s) that may affect neuromuscular block and/or trial assessments.
* Are dialysis-dependent or have severe renal insufficiency (defined as estimated creatinine clearance of <30 mL/min.).
* Have or are suspected of having a personal history or family history (parents, grandparents, or siblings) of malignant hyperthermia.
* Have or are suspected of having an allergy (e.g., hypersensitivity and/or anaphylactic reaction) to study treatments or its/their excipients, to opioids/opiates, muscle relaxants or their excipients, or other medication(s) used during general anesthesia.
* Have received or are planning to receive toremifene within 24 hours before or within 24 hours after study medication administration.
* Have any condition that would contraindicate the administration of study medication.
* Are currently pregnant, attempting to become pregnant, or lactating.
* Have any clinically significant condition or situation (e.g., anatomical malformation that complicates intubation) other than the condition being studied that, in the opinion of the investigator, would interfere with the trial evaluations or optimal participation in the trial.
* Are currently participating in or has participated in an interventional clinical trial with an investigational compound (including any other current or ongoing trial with a Sugammadex treatment arm) or device within 30 days of signing the informed consent form of this current trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-29 (Actual); Study Completion 2019-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (24):
- United States (13):
  - University California / Davis ( Site 2001), Sacramento, California
  - Jackson Memorial Hospital/University of Miami ( Site 2007), Miami, Florida
  - University of Kansas Medical Center ( Site 2049), Kansas City, Kansas
  - William Beaumont Hospital - Royal Oak ( Site 2033), Royal Oak, Michigan
  - University Hospital- Columbia MO ( Site 2060), Columbia, Missouri
  - Robert Wood Johnson University Hospital ( Site 2037), New Brunswick, New Jersey
  - Mission Hospital - St. Joseph ( Site 2015), Asheville, North Carolina
  - Cleveland Clinic Foundation ( Site 2031), Cleveland, Ohio
  - Temple University Hospital ( Site 2004), Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center ( Site 2032), Nashville, Tennessee
  - Hermann Drive Surgical Center ( Site 2020), Houston, Texas
  - Hermann Drive Surgical Center ( Site 2059), Houston, Texas
  - Zablocki VA Medical Center ( Site 2011), Milwaukee, Wisconsin
- Sozialmedizinisches Zentrum Ost - Donauspital ( Site 2150), Vienna, Austria
- Universitaire Ziekenhuis Antwerpen - UZA ( Site 2200), Edegem, Belgium
- Denmark (2):
  - Rigshospitalet ( Site 2253), Copenhagen
  - Bispebjerg og Frederiksberg Hospital ( Site 2250), Copenhagen NV
- Germany (7):
  - Johanniter Krankenhaus Bonn ( Site 2353), Bonn
  - Diakovere Annastift gGmbH ( Site 2355), Hanover
  - Universitatsklinikum Giessen und Marburg GmbH ( Site 2356), Marburg
  - Klinikum Rechts der Isar Technische Universitaet Muenchen ( Site 2350), München
  - St. Franziskus-Hospital ( Site 2354), Münster
  - Klinikum am Steinenberg Reutlingen ( Site 2352), Reutlingen
  - Josephs-Hospitals Warendorf ( Site 2351), Warendorf

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Mostoller K, Wrishko R, Maganti L, Herring WJ, van Zutphen-van Geffen M. Pharmacokinetics of Sugammadex Dosed by Actual and Ideal Body Weight in Patients With Morbid Obesity Undergoing Surgery. Clin Transl Sci. 2021 Mar;14(2):737-744. doi: 10.1111/cts.12941. Epub 2020 Dec 16. PMID 33278332
- [Derived] Horrow JC, Li W, Blobner M, Lombard J, Speek M, DeAngelis M, Herring WJ. Actual versus ideal body weight dosing of sugammadex in morbidly obese patients offers faster reversal of rocuronium- or vecuronium-induced deep or moderate neuromuscular block: a randomized clinical trial. BMC Anesthesiol. 2021 Feb 27;21(1):62. doi: 10.1186/s12871-021-01278-w. PMID 33639839

RESULTS

PARTICIPANT FLOW:
Groups:
- Sugammadex 2 mg/kg Actual Body Weight (ABW): Following administration of NMBA, participants received a single intravenous (i.v.) bolus of Sugammadex at 2 mg/kg as determined utilizing participant ABW. A treatment dose of 2 mg/kg was used for reversal of moderate NMB.
- Sugammadex 2 mg/kg Ideal Body Weight (IBW): Following administration of NMBA, participants received a single i.v. bolus of Sugammadex at 2 mg/kg as determined utilizing participant IBW. A treatment dose of 2 mg/kg was used for reversal of moderate NMB.
Period: Overall Study
Arm/Group | Sugammadex 2 mg/kg Actual Body Weight (ABW) | Sugammadex 4 mg/kg ABW | Sugammadex 2 mg/kg Ideal Body Weight (IBW) | Sugammadex 4 mg/kg IBW | Neostigmine/Glycopyrrolate
Started | 41 | 41 | 41 | 42 | 42
Treated | 38 | 38 | 38 | 36 | 38
Completed | 38 | 37 | 37 | 36 | 37
Not Completed | 3 | 4 | 4 | 6 | 5
Not completed — Death | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 2 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1 | 0
Not completed — Study medication not received as planned | 2 | 3 | 2 | 3 | 2
Not completed — Screen Failure | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Sugammadex 2 mg/kg ABW: Following administration of NMBA, participants received a single i.v. bolus of Sugammadex at 2 mg/kg as determined utilizing participant ABW. A treatment dose of 2 mg/kg was used for reversal of moderate NMB.
- Total: Total of all reporting groups
Arm/Group | Sugammadex 2 mg/kg ABW | Sugammadex 4 mg/kg ABW | Sugammadex 2 mg/kg IBW | Sugammadex 4 mg/kg IBW | Neostigmine/Glycopyrrolate | Total
Number analyzed (Participants) | 41 | 41 | 41 | 42 | 42 | 207
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.7 (14.4) | 46.4 (11.2) | 47.6 (14.5) | 49.2 (11.7) | 47.7 (13.3) | 47.7 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 24 | 30 | 32 | 29 | 149
  Male | 7 | 17 | 11 | 10 | 13 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 1 | 5 | 2 | 13
  Not Hispanic or Latino | 38 | 37 | 40 | 37 | 39 | 191
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 2 | 2 | 4 | 3 | 3 | 14
  White | 39 | 39 | 37 | 38 | 38 | 191
  More than one race | 0 | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Recovery (TTR) of Participant Train Of Four (TOF) Ratio to ≥0.9: Primary Kaplan-Meier Analysis
Description: The primary efficacy analysis of TTR of TOF ratio to ≥0.9 was performed by estimating event rates within each treatment group using the Kaplan-Meier method. TTR was monitored by applying electrical stimulations to the ulnar nerve every 15 seconds and assessing twitch response at the adductor pollicis muscle. T1 and T4 refer to magnitudes of the first and fourth twitches respectively, after nerve stimulation. The T4/T1 ratio (TOF; expressed as a decimal of up to 1.0) indicates the extent of recovery from NMB. A faster TTR of the TOF ratio to 0.9 indicates faster recovery from NMB. As specified by the protocol, analyses for this outcome measure were conducted in participants pooled by dosing method across depth of NMB (Sugammadex ABW [2 mg/kg ABW plus 4 mg/kg ABW] and Sugammadex IBW [2 mg/kg IBW plus 4 mg/kg IBW]) as well as in all randomized treatment arms separated by depth of NMB (Sugammadex 2 mg/kg ABW, Sugammadex 4 mg/kg ABW, Sugammadex 2 mg/kg IBW, and Sugammadex 4 mg/kg IBW).
Time Frame: Up to 76 minutes
Population: All randomized participants dosed with both an NMBA and an NMB reversal agent (study treatment) with ≥1 post-randomization efficacy assessment. As specified by the protocol, analysis was performed in treatment arms pooled by dosing method across depth of NMB as well as in all randomized treatment arms separated by depth of NMB.
Measure: Median (95% Confidence Interval); unit: Minutes
Groups:
- Sugammadex ABW (2 mg/kg ABW Plus 4 mg/kg ABW): Following administration of NMBA, participants who received a single i.v. bolus of Sugammadex at 2 mg/kg as determined utilizing participant ABW, and those who received a single i.v. bolus of Sugammadex at 4 mg/kg as determined utilizing participant ABW were pooled by dosing method across depth of NMB. Treatment doses of 2 mg/kg and 4 mg/kg were used for reversal of moderate NMB and deep NMB respectively.
- Sugammadex IBW (2 mg/kg IBW Plus 4 mg/kg IBW): Following administration of NMBA, participants who received a single i.v. bolus of Sugammadex at 2 mg/kg as determined utilizing participant IBW, and those who received a single i.v. bolus of Sugammadex at 4 mg/kg as determined utilizing participant IBW were pooled by dosing method across depth of NMB. Treatment doses of 2 mg/kg and 4 mg/kg were used for reversal of moderate NMB and deep NMB respectively.
Arm/Group | Sugammadex 2 mg/kg ABW | Sugammadex 4 mg/kg ABW | Sugammadex ABW (2 mg/kg ABW Plus 4 mg/kg ABW) | Sugammadex 2 mg/kg IBW | Sugammadex 4 mg/kg IBW | Sugammadex IBW (2 mg/kg IBW Plus 4 mg/kg IBW) | Neostigmine/Glycopyrrolate
Number analyzed (Participants) | 38 | 37 | 75 | 37 | 36 | 73 | 38
Minutes | 1.7 [1.5 to 2.1] | 1.8 [1.5 to 2.1] | 1.8 [1.6 to 2.1] | 3.4 [2.2 to 4.4] | 3.3 [2.4 to 4.2] | 3.3 [2.6 to 4.1] | 34.5 [27.0 to 67.4]
Statistical Analysis 1: Comparison: Sugammadex 2 mg/kg ABW vs Sugammadex 2 mg/kg IBW; Test type: Superiority; p = 0.0075, Log Rank; Hazard Ratio (HR) = 1.92, 95% CI 2-sided [1.18 to 3.10] — Cox regression model
Statistical Analysis 2: Comparison: Sugammadex 2 mg/kg ABW vs Neostigmine/Glycopyrrolate; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 25.90, 95% CI 2-sided [9.72 to 69.03] — Cox regression model
Statistical Analysis 3: Comparison: Sugammadex 2 mg/kg IBW vs Neostigmine/Glycopyrrolate; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 61.40, 95% CI 2-sided [14.13 to 266.77] — Cox regression model
Statistical Analysis 4: Comparison: Sugammadex 4 mg/kg ABW vs Sugammadex 4 mg/kg IBW; Test type: Superiority; p = 0.0005, Log Rank; Hazard Ratio (HR) = 2.38, 95% CI 2-sided [1.44 to 3.93] — Cox regression model
Statistical Analysis 5: Comparison: Sugammadex ABW (2 mg/kg ABW Plus 4 mg/kg ABW) vs Sugammadex IBW (2 mg/kg IBW Plus 4 mg/kg IBW); Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 2.13, 95% CI 2-sided [1.50 to 3.01] — Cox regression model

2. Primary Outcome: Percentage of Participants With Treatment-Emergent Sinus Bradycardia Events
Description: The percentage of participants experiencing treatment-emergent bradycardia events were identified with continuous electrocardiogram (ECG) monitoring. Treatment-emergent sinus bradycardia is defined as a heart rate <60 bpm that has also decreased more than 20% compared to participant baseline heart rate value, sustained for at least 1 minute after administration of study intervention. Treatment-emergent sinus bradycardia events may or may not be considered an adverse event (AE), as determined by investigator judgment. As specified by the protocol, analyses for this outcome measure were conducted in participants pooled by dosing method across depth of NMB (Sugammadex ABW [2 mg/kg ABW plus 4 mg/kg ABW] and Sugammadex IBW [2 mg/kg IBW plus 4 mg/kg IBW]) as well as in all randomized treatment arms separated by depth of NMB (Sugammadex 2 mg/kg ABW, Sugammadex 4 mg/kg ABW, Sugammadex 2 mg/kg IBW, and Sugammadex 4 mg/kg IBW).
Time Frame: Up to 35 minutes
Population: All randomized participants who received at least one dose of study treatment. As specified by the protocol, analysis was performed in treatment arms pooled by dosing method across depth of NMB as well as in all randomized treatment arms separated by depth of NMB.
Measure: Number; unit: Percentage of participants
Arm/Group | Sugammadex 2 mg/kg ABW | Sugammadex 4 mg/kg ABW | Sugammadex ABW (2 mg/kg ABW Plus 4 mg/kg ABW) | Sugammadex 2 mg/kg IBW | Sugammadex 4 mg/kg IBW | Sugammadex IBW (2 mg/kg IBW Plus 4 mg/kg IBW) | Neostigmine/Glycopyrrolate
Number analyzed (Participants) | 38 | 38 | 76 | 38 | 36 | 74 | 38
Percentage of participants | 5.3 | 5.3 | 5.3 | 2.6 | 5.6 | 4.1 | 2.6
Statistical Analysis 1: Comparison: Sugammadex 2 mg/kg ABW vs Sugammadex 2 mg/kg IBW; Test type: Superiority; p = 0.602, Miettinen & Nurminen method; Difference in percentage = 2.3, 95% CI 2-sided [-9.6 to 15.0]
Statistical Analysis 2: Comparison: Sugammadex 4 mg/kg ABW vs Sugammadex 4 mg/kg IBW; Test type: Superiority; p = 0.969, Miettinen & Nurminen method; Difference in percentage = 0.2, 95% CI 2-sided [-13.4 to 13.5]
Statistical Analysis 3: Comparison: Sugammadex 2 mg/kg ABW vs Neostigmine/Glycopyrrolate; Test type: Superiority; p = 0.567, Miettinen & Nurminen method; Difference in percentage = 2.6, 95% CI 2-sided [-8.7 to 15.0]
Statistical Analysis 4: Comparison: Sugammadex 4 mg/kg ABW vs Neostigmine/Glycopyrrolate; Test type: Superiority; p = 0.571, Miettinen & Nurminen method; Difference in percentage = 2.6, 95% CI 2-sided [-8.8 to 15.0]
Statistical Analysis 5: Comparison: Sugammadex 2 mg/kg IBW vs Neostigmine/Glycopyrrolate; Test type: Superiority; p = 0.950, Miettinen & Nurminen method; Difference in percentage = -0.2, 95% CI 2-sided [-11.6 to 10.9]
Statistical Analysis 6: Comparison: Sugammadex 4 mg/kg IBW vs Neostigmine/Glycopyrrolate; Test type: Superiority; p = 0.528, Miettinen & Nurminen method; Difference in percentage = 2.9, 95% CI 2-sided [-8.4 to 15.9]
Statistical Analysis 7: Comparison: Sugammadex ABW (2 mg/kg ABW Plus 4 mg/kg ABW) vs Sugammadex IBW (2 mg/kg IBW Plus 4 mg/kg IBW); Test type: Superiority; p = 0.709, Miettinen & Nurminen method; Difference in percentage = 1.3, 95% CI 2-sided [-6.8 to 9.6]

3. Primary Outcome: Percentage of Participants With Treatment-Emergent Sinus Tachycardia Events
Description: The percentage of participants experiencing treatment-emergent sinus tachycardia events were identified with continuous ECG monitoring. Treatment-emergent sinus tachycardia is defined as a heart rate ≥100 bpm that has also increased more than 20% compared to participant baseline heart rate value, sustained for at least 1 minute after administration of study intervention. Treatment-emergent sinus tachycardia events may or may not be considered an AE, as determined by investigator judgment. As specified by the protocol, analyses for this outcome measure were conducted in participants pooled by dosing method across depth of NMB (Sugammadex ABW [2 mg/kg ABW plus 4 mg/kg ABW] and Sugammadex IBW [2 mg/kg IBW plus 4 mg/kg IBW]) as well as in all randomized treatment arms separated by depth of NMB (Sugammadex 2 mg/kg ABW, Sugammadex 4 mg/kg ABW, Sugammadex 2 mg/kg IBW, and Sugammadex 4 mg/kg IBW).
Time Frame: Up to 35 minutes
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Sugammadex 2 mg/kg ABW | Sugammadex 4 mg/kg ABW | Sugammadex ABW (2 mg/kg ABW Plus 4 mg/kg ABW) | Sugammadex 2 mg/kg IBW | Sugammadex 4 mg/kg IBW | Sugammadex IBW (2 mg/kg IBW Plus 4 mg/kg IBW) | Neostigmine/Glycopyrrolate
Number analyzed (Participants) | 38 | 38 | 76 | 38 | 36 | 74 | 38
Percentage of participants | 10.5 | 13.2 | 11.8 | 7.9 | 2.8 | 5.4 | 7.9
Statistical Analysis 1: Comparison: Sugammadex 2 mg/kg ABW vs Sugammadex 2 mg/kg IBW; Test type: Superiority; p = 0.738, Miettinen & Nurminen method; Difference in percentage = 2.2, 95% CI 2-sided [-12.3 to 17.4]
Statistical Analysis 2: Comparison: Sugammadex 4 mg/kg ABW vs Sugammadex 4 mg/kg IBW; Test type: Superiority; p = 0.077, Miettinen & Nurminen method; Difference in percentage = 11.1, 95% CI 2-sided [-1.7 to 26.3]
Statistical Analysis 3: Comparison: Sugammadex 2 mg/kg ABW vs Neostigmine/Glycopyrrolate; Test type: Superiority; p = 0.717, Miettinen & Nurminen method; Difference in percentage = 2.4, 95% CI 2-sided [-12.0 to 16.4]
Statistical Analysis 4: Comparison: Sugammadex 4 mg/kg ABW vs Neostigmine/Glycopyrrolate; Test type: Superiority; p = 0.486, Miettinen & Nurminen method; Difference in percentage = 5.0, 95% CI 2-sided [-9.9 to 19.7]
Statistical Analysis 5: Comparison: Sugammadex 2 mg/kg IBW vs Neostigmine/Glycopyrrolate; Test type: Superiority; p = 0.849, Miettinen & Nurminen method; Difference in percentage = -1.2, 95% CI 2-sided [-16.2 to 12.4]
Statistical Analysis 6: Comparison: Sugammadex 4 mg/kg IBW vs Neostigmine/Glycopyrrolate; Test type: Superiority; p = 0.339, Miettinen & Nurminen method; Difference in percentage = -4.9, 95% CI 2-sided [-18.2 to 6.7]
Statistical Analysis 7: Comparison: Sugammadex ABW (2 mg/kg ABW Plus 4 mg/kg ABW) vs Sugammadex IBW (2 mg/kg IBW Plus 4 mg/kg IBW); Test type: Superiority; p = 0.149, Miettinen & Nurminen method; Difference in percentage = 6.6, 95% CI 2-sided [-2.6 to 16.8]

4. Primary Outcome: Percentage of Participants With Other Treatment-Emergent Cardiac Arrhythmia Events
Description: The percentage of participants experiencing other treatment-emergent cardiac arrhythmia events were identified with continuous ECG monitoring. Other treatment-emergent cardiac arrhythmias are defined as new or worsening arrhythmias (e.g., atrial fibrillation, atrial tachyarrhythmia, ventricular fibrillation, or ventricular tachyarrhythmia), sustained for at least 1 minute after administration of study intervention. Worsening arrhythmia events may or may not be considered an AE, as determined by investigator judgment. As specified by the protocol, analyses for this outcome measure were conducted in participants pooled by dosing method across depth of NMB (Sugammadex ABW [2 mg/kg ABW plus 4 mg/kg ABW] and Sugammadex IBW [2 mg/kg IBW plus 4 mg/kg IBW]) as well as in all randomized treatment arms separated by depth of NMB (Sugammadex 2 mg/kg ABW, Sugammadex 4 mg/kg ABW, Sugammadex 2 mg/kg IBW, and Sugammadex 4 mg/kg IBW).
Time Frame: Up to 35 minutes
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Sugammadex 2 mg/kg ABW | Sugammadex 4 mg/kg ABW | Sugammadex ABW (2 mg/kg ABW Plus 4 mg/kg ABW) | Sugammadex 2 mg/kg IBW | Sugammadex 4 mg/kg IBW | Sugammadex IBW (2 mg/kg IBW Plus 4 mg/kg IBW) | Neostigmine/Glycopyrrolate
Number analyzed (Participants) | 38 | 38 | 76 | 38 | 36 | 74 | 38
Percentage of participants | 0.0 | 0.0 | 0.0 | 2.6 | 0.0 | 1.4 | 2.6
Statistical Analysis 1: Comparison: Sugammadex 2 mg/kg ABW vs Sugammadex 2 mg/kg IBW; Test type: Superiority; p = 0.299, Miettinen & Nurminen method; Difference in percentage = -2.7, 95% CI 2-sided [-13.9 to 6.7]
Statistical Analysis 2: Comparison: Sugammadex 4 mg/kg ABW vs Sugammadex 4 mg/kg IBW; Test type: Superiority; p > 0.999, Miettinen & Nurminen method; Difference in percentage = 0.0, 95% CI 2-sided [-9.9 to 9.4]
Statistical Analysis 3: Comparison: Sugammadex 2 mg/kg ABW vs Neostigmine/Glycopyrrolate; Test type: Superiority; p = 0.326, Miettinen & Nurminen method; Difference in percentage = -2.6, 95% CI 2-sided [-13.7 to 7.0]
Statistical Analysis 4: Comparison: Sugammadex 4 mg/kg ABW vs Neostigmine/Glycopyrrolate; Test type: Superiority; p = 0.335, Miettinen & Nurminen method; Difference in percentage = -2.5, 95% CI 2-sided [-13.6 to 7.1]
Statistical Analysis 5: Comparison: Sugammadex 2 mg/kg IBW vs Neostigmine/Glycopyrrolate; Test type: Superiority; p = 0.935, Miettinen & Nurminen method; Difference in percentage = 0.3, 95% CI 2-sided [-11.1 to 11.9]
Statistical Analysis 6: Comparison: Sugammadex 4 mg/kg IBW vs Neostigmine/Glycopyrrolate; Test type: Superiority; p = 0.326, Miettinen & Nurminen method; Difference in percentage = -2.7, 95% CI 2-sided [-13.8 to 7.3]
Statistical Analysis 7: Comparison: Sugammadex ABW (2 mg/kg ABW Plus 4 mg/kg ABW) vs Sugammadex IBW (2 mg/kg IBW Plus 4 mg/kg IBW); Test type: Superiority; p = 0.299, Miettinen & Nurminen method; Difference in percentage = -1.4, 95% CI 2-sided [-7.5 to 3.5]

5. Primary Outcome: Percentage of Participants Experiencing an Adverse Event (AE) After Administration of Study Intervention
Description: The percentage of participants experiencing an AE following administration of study intervention was monitored. An AE is any unfavorable and unintended medical occurrence, symptom, or disease witnessed in a participant, regardless of whether or not a causal relationship with the study treatment can be demonstrated. Further, any worsening (i.e. any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of the study treatment is also considered an AE. As specified by the protocol, analyses for this outcome measure were conducted in participants pooled by dosing method across depth of NMB (Sugammadex ABW [2 mg/kg ABW plus 4 mg/kg ABW] and Sugammadex IBW [2 mg/kg IBW plus 4 mg/kg IBW]) as well as in all randomized treatment arms separated by depth of NMB (Sugammadex 2 mg/kg ABW, Sugammadex 4 mg/kg ABW, Sugammadex 2 mg/kg IBW, and Sugammadex 4 mg/kg IBW).
Time Frame: Up to 7 days
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Sugammadex 2 mg/kg ABW | Sugammadex 4 mg/kg ABW | Sugammadex ABW (2 mg/kg ABW Plus 4 mg/kg ABW) | Sugammadex 2 mg/kg IBW | Sugammadex 4 mg/kg IBW | Sugammadex IBW (2 mg/kg IBW Plus 4 mg/kg IBW) | Neostigmine/Glycopyrrolate
Number analyzed (Participants) | 38 | 38 | 76 | 38 | 36 | 74 | 38
Percentage of participants | 94.7 | 86.8 | 90.8 | 94.7 | 91.7 | 93.2 | 89.5
Statistical Analysis 1: Comparison: Sugammadex 2 mg/kg ABW vs Sugammadex 2 mg/kg IBW; Test type: Superiority; Difference in percentage = 0.1, 95% CI 2-sided [-12.7 to 13.1] — Miettinen and Nurminen method
Statistical Analysis 2: Comparison: Sugammadex 4 mg/kg ABW vs Sugammadex 4 mg/kg IBW; Test type: Superiority; Difference in percentage = -3.6, 95% CI 2-sided [-19.6 to 12.2] — Miettinen and Nurminen method
Statistical Analysis 3: Comparison: Sugammadex 2 mg/kg ABW vs Neostigmine/Glycopyrrolate; Test type: Superiority; Difference in percentage = 5.1, 95% CI 2-sided [-8.1 to 19.7] — Miettinen and Nurminen method
Statistical Analysis 4: Comparison: Sugammadex 4 mg/kg ABW vs Neostigmine/Glycopyrrolate; Test type: Superiority; Difference in percentage = -2.6, 95% CI 2-sided [-18.0 to 13.1] — Miettinen and Nurminen method
Statistical Analysis 5: Comparison: Sugammadex 2 mg/kg IBW vs Neostigmine/Glycopyrrolate; Test type: Superiority; Difference in percentage = 4.4, 95% CI 2-sided [-9.6 to 19.2] — Miettinen and Nurminen method
Statistical Analysis 6: Comparison: Sugammadex 4 mg/kg IBW vs Neostigmine/Glycopyrrolate; Test type: Superiority; Difference in percentage = 2.2, 95% CI 2-sided [-12.5 to 17.0] — Miettinen and Nurminen method
Statistical Analysis 7: Comparison: Sugammadex ABW (2 mg/kg ABW Plus 4 mg/kg ABW) vs Sugammadex IBW (2 mg/kg IBW Plus 4 mg/kg IBW); Test type: Superiority; Difference in percentage = -1.8, 95% CI 2-sided [-11.4 to 7.8] — Miettinen and Nurminen method

6. Primary Outcome: Percentage of Participants Experiencing a Serious Adverse Event (SAE) After Administration of Study Intervention
Description: The percentage of participants experiencing an SAE following administration of study intervention was monitored. An SAE is an adverse event that: results in death; is life threatening; results in persistent or significant disability or incapacity; results in or prolongs a hospitalization; is a congenital anomaly or birth defect; is a cancer; or may jeopardize the participant, potentially requiring medical or surgical intervention. As specified by the protocol, analyses for this outcome measure were conducted in participants pooled by dosing method across depth of NMB (Sugammadex ABW [2 mg/kg ABW plus 4 mg/kg ABW] and Sugammadex IBW [2 mg/kg IBW plus 4 mg/kg IBW]) as well as in all randomized treatment arms separated by depth of NMB (Sugammadex 2 mg/kg ABW, Sugammadex 4 mg/kg ABW, Sugammadex 2 mg/kg IBW, and Sugammadex 4 mg/kg IBW).
Time Frame: Up to 7 days
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Sugammadex 2 mg/kg ABW | Sugammadex 4 mg/kg ABW | Sugammadex ABW (2 mg/kg ABW Plus 4 mg/kg ABW) | Sugammadex 2 mg/kg IBW | Sugammadex 4 mg/kg IBW | Sugammadex IBW (2 mg/kg IBW Plus 4 mg/kg IBW) | Neostigmine/Glycopyrrolate
Number analyzed (Participants) | 38 | 38 | 76 | 38 | 36 | 74 | 38
Percentage of participants | 2.6 | 0.0 | 1.3 | 5.3 | 8.3 | 6.8 | 7.9
Statistical Analysis 1: Comparison: Sugammadex 2 mg/kg ABW vs Sugammadex 2 mg/kg IBW; Test type: Superiority; Difference in percentage = -2.6, 95% CI 2-sided [-15.2 to 9.1] — Miettinen and Nurminen method
Statistical Analysis 2: Comparison: Sugammadex 4 mg/kg ABW vs Sugammadex 4 mg/kg IBW; Test type: Superiority; Difference in percentage = -8.5, 95% CI 2-sided [-22.3 to 1.3] — Miettinen and Nurminen method
Statistical Analysis 3: Comparison: Sugammadex 2 mg/kg ABW vs Neostigmine/Glycopyrrolate; Test type: Superiority; Difference in percentage = -5.3, 95% CI 2-sided [-18.8 to 6.8] — Miettinen and Nurminen method
Statistical Analysis 4: Comparison: Sugammadex 4 mg/kg ABW vs Neostigmine/Glycopyrrolate; Test type: Superiority; Difference in percentage = -8.0, 95% CI 2-sided [-21.2 to 1.8] — Miettinen and Nurminen method
Statistical Analysis 5: Comparison: Sugammadex 2 mg/kg IBW vs Neostigmine/Glycopyrrolate; Test type: Superiority; Difference in percentage = -2.9, 95% CI 2-sided [-17.0 to 10.5] — Miettinen and Nurminen method
Statistical Analysis 6: Comparison: Sugammadex 4 mg/kg IBW vs Neostigmine/Glycopyrrolate; Test type: Superiority; Difference in percentage = 0.5, 95% CI 2-sided [-14.0 to 15.5] — Miettinen and Nurminen method
Statistical Analysis 7: Comparison: Sugammadex ABW (2 mg/kg ABW Plus 4 mg/kg ABW) vs Sugammadex IBW (2 mg/kg IBW Plus 4 mg/kg IBW); Test type: Superiority; Difference in percentage = -5.5, 95% CI 2-sided [-13.9 to 1.2] — Miettinen and Nurminen method

7. Primary Outcome: Percentage of Participants Experiencing an Event of Clinical Interest (ECI) After Administration of Study Intervention
Description: The percentage of participants experiencing an ECI following administration of study intervention was monitored. ECIs are a discrete set of both AEs and SAEs, specifically designated as such for the trial. For the purposes of this investigation, ECIs included 1) drug-induced liver injury; 2) clinically-relevant arrhythmias, inclusive of bradycardia and tachycardia defined as events necessitating intervention, as determined by investigator judgment; and 3) instances of hypersensitivity and/or anaphylaxis adjudicated by an external expert Adjudication Committee. As specified by the protocol, analyses for this outcome measure were conducted in participants pooled by dosing method across depth of NMB (Sugammadex ABW [2 mg/kg ABW plus 4 mg/kg ABW] and Sugammadex IBW [2 mg/kg IBW plus 4 mg/kg IBW]) as well as in all randomized treatment arms separated by depth of NMB (Sugammadex 2 mg/kg ABW, Sugammadex 4 mg/kg ABW, Sugammadex 2 mg/kg IBW, and Sugammadex 4 mg/kg IBW).
Time Frame: Up to 7 days
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Sugammadex 2 mg/kg ABW | Sugammadex 4 mg/kg ABW | Sugammadex ABW (2 mg/kg ABW Plus 4 mg/kg ABW) | Sugammadex 2 mg/kg IBW | Sugammadex 4 mg/kg IBW | Sugammadex IBW (2 mg/kg IBW Plus 4 mg/kg IBW) | Neostigmine/Glycopyrrolate
Number analyzed (Participants) | 38 | 38 | 76 | 38 | 36 | 74 | 38
Percentage of participants | 0.0 | 2.6 | 1.3 | 2.6 | 2.8 | 2.7 | 2.6
Statistical Analysis 1: Comparison: Sugammadex 2 mg/kg ABW vs Sugammadex 2 mg/kg IBW; Test type: Superiority; Difference in percentage = -2.4, 95% CI 2-sided [-13.4 to 7.3] — Miettinen and Nurminen method
Statistical Analysis 2: Comparison: Sugammadex 4 mg/kg ABW vs Sugammadex 4 mg/kg IBW; Test type: Superiority; Difference in percentage = -0.4, 95% CI 2-sided [-12.3 to 10.8] — Miettinen and Nurminen method
Statistical Analysis 3: Comparison: Sugammadex 2 mg/kg ABW vs Neostigmine/Glycopyrrolate; Test type: Superiority; Difference in percentage = -2.6, 95% CI 2-sided [-13.7 to 7.0] — Miettinen and Nurminen method
Statistical Analysis 4: Comparison: Sugammadex 4 mg/kg ABW vs Neostigmine/Glycopyrrolate; Test type: Superiority; Difference in percentage = 0.2, 95% CI 2-sided [-11.2 to 11.7] — Miettinen and Nurminen method
Statistical Analysis 5: Comparison: Sugammadex 2 mg/kg IBW vs Neostigmine/Glycopyrrolate; Test type: Superiority; Difference in percentage = -0.2, 95% CI 2-sided [-11.5 to 11.0] — Miettinen and Nurminen method
Statistical Analysis 6: Comparison: Sugammadex 4 mg/kg IBW vs Neostigmine/Glycopyrrolate; Test type: Superiority; Difference in percentage = 0.2, 95% CI 2-sided [-11.0 to 12.0] — Miettinen and Nurminen method

8. Secondary Outcome: Percentage of Participants With Prolonged (>10 Minutes) Time to Recovery (TTR) of the Train Of Four (TOF) Ratio to ≥0.9
Description: Following administration of study intervention, the percentage of participants experiencing prolonged (>10 minutes) recovery to a TOF ratio ≥0.9 was calculated. TTR was monitored by applying electrical stimulations to the ulnar nerve every 15 seconds and assessing twitch response at the adductor pollicis muscle. T1 and T4 refer to magnitudes of the first and fourth twitches respectively, after nerve stimulation. The T4/T1 ratio (TOF; expressed as a decimal of up to 1.0) indicates the extent of recovery from NMB. A faster TTR of the TOF ratio to 0.9 indicates faster recovery from NMB. As specified by the protocol, analyses for this outcome measure were conducted in participants pooled by dosing method across depth of NMB (Sugammadex ABW [2 mg/kg ABW plus 4 mg/kg ABW] and Sugammadex IBW [2 mg/kg IBW plus 4 mg/kg IBW]) as well as in all randomized treatment arms separated by depth of NMB (Sugammadex 2 mg/kg ABW, Sugammadex 4 mg/kg ABW, Sugammadex 2 mg/kg IBW, and Sugammadex 4 mg/kg IBW).
Time Frame: Up to 76 minutes
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Sugammadex 2 mg/kg ABW | Sugammadex 4 mg/kg ABW | Sugammadex ABW (2 mg/kg ABW Plus 4 mg/kg ABW) | Sugammadex 2 mg/kg IBW | Sugammadex 4 mg/kg IBW | Sugammadex IBW (2 mg/kg IBW Plus 4 mg/kg IBW) | Neostigmine/Glycopyrrolate
Number analyzed (Participants) | 38 | 37 | 75 | 37 | 36 | 73 | 38
Percentage of participants | 7.9 | 2.7 | 5.3 | 5.4 | 0.0 | 2.7 | 84.2
Statistical Analysis 1: Comparison: Sugammadex 2 mg/kg ABW vs Sugammadex 2 mg/kg IBW; Test type: Superiority; Difference in percentage = 3.0, 95% CI 2-sided [-10.8 to 16.9] — Miettinen and Nurminen method
Statistical Analysis 2: Comparison: Sugammadex 2 mg/kg ABW vs Neostigmine/Glycopyrrolate; Test type: Superiority; Difference in percentage = -76.1, 95% CI 2-sided [-87.2 to -57.6] — Miettinen and Nurminen method
Statistical Analysis 3: Comparison: Sugammadex 2 mg/kg IBW vs Neostigmine/Glycopyrrolate; Test type: Superiority; Difference in percentage = -78.7, 95% CI 2-sided [-88.8 to -61.1] — Miettinen and Nurminen method
Statistical Analysis 4: Comparison: Sugammadex 4 mg/kg ABW vs Sugammadex 4 mg/kg IBW; Test type: Superiority; Difference in percentage = 2.8, 95% CI 2-sided [-7.2 to 14.2] — Miettinen and Nurminen method
Statistical Analysis 5: Comparison: Sugammadex ABW (2 mg/kg ABW Plus 4 mg/kg ABW) vs Sugammadex IBW (2 mg/kg IBW Plus 4 mg/kg IBW); Test type: Superiority; Difference in percentage = 2.9, 95% CI 2-sided [-4.8 to 11.0] — Miettinen and Nurminen method

9. Secondary Outcome: Time to Recovery (TTR) of Participant Train of Four (TOF) Ratio to ≥0.9: Secondary Geometric Mean Analysis
Description: The secondary efficacy analysis of TTR of participant TOF ratio to ≥0.9 was performed by estimating the geometric mean of TTR within each treatment group. TTR was monitored by applying electrical stimulations to the ulnar nerve every 15 seconds and assessing twitch response at the adductor pollicis muscle. T1 and T4 refer to magnitudes of the first and fourth twitches respectively, after nerve stimulation. The T4/T1 ratio (TOF; expressed as a decimal of up to 1.0) indicates the extent of recovery from NMB. A faster TTR of the TOF ratio to 0.9 indicates faster recovery from NMB. As specified by the protocol, analyses for this outcome measure were conducted in participants pooled by dosing method across depth of NMB (Sugammadex ABW [2 mg/kg ABW plus 4 mg/kg ABW] and Sugammadex IBW [2 mg/kg IBW plus 4 mg/kg IBW]) as well as in all randomized treatment arms separated by depth of NMB (Sugammadex 2 mg/kg ABW, Sugammadex 4 mg/kg ABW, Sugammadex 2 mg/kg IBW, and Sugammadex 4 mg/kg IBW).
Time Frame: Up to 76 minutes
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Sugammadex 2 mg/kg ABW | Sugammadex 4 mg/kg ABW | Sugammadex ABW (2 mg/kg ABW Plus 4 mg/kg ABW) | Sugammadex 2 mg/kg IBW | Sugammadex 4 mg/kg IBW | Sugammadex IBW (2 mg/kg IBW Plus 4 mg/kg IBW) | Neostigmine/Glycopyrrolate
Number analyzed (Participants) | 38 | 37 | 75 | 37 | 36 | 73 | 38
Minutes | 2.0 [1.7 to 2.5] | 1.9 [1.5 to 2.3] | 2.0 [1.7 to 2.3] | 3.2 [2.6 to 3.9] | 3.5 [2.9 to 4.3] | 3.3 [2.9 to 3.8] | 23.1 [18.3 to 29.2]
Statistical Analysis 1: Comparison: Sugammadex 2 mg/kg ABW vs Sugammadex 2 mg/kg IBW; Test type: Superiority; Ratio of geometric means = 0.64, 95% CI 2-sided [0.48 to 0.86] — Log transformation and t-distribution
Statistical Analysis 2: Comparison: Sugammadex 2 mg/kg ABW vs Neostigmine/Glycopyrrolate; Test type: Superiority; Ratio of geometric means = 0.09, 95% CI 2-sided [0.06 to 0.12] — Log transformation and t-distribution
Statistical Analysis 3: Comparison: Sugammadex 2 mg/kg IBW vs Neostigmine/Glycopyrrolate; Test type: Superiority; Ratio of geometric means = 0.14, 95% CI 2-sided [0.10 to 0.19] — Log transformation and t-distribution
Statistical Analysis 4: Comparison: Sugammadex 4 mg/kg ABW vs Sugammadex 4 mg/kg IBW; Test type: Superiority; Ratio of geometric means = 0.54, 95% CI 2-sided [0.40 to 0.71] — Log transformation and t-distribution
Statistical Analysis 5: Comparison: Sugammadex ABW (2 mg/kg ABW Plus 4 mg/kg ABW) vs Sugammadex IBW (2 mg/kg IBW Plus 4 mg/kg IBW); Test type: Superiority; Ratio of geometric means = 0.59, 95% CI 2-sided [0.48 to 0.72] — Log transformation and t-distribution

10. Secondary Outcome: Time to Recovery (TTR) of Participant Train of Four (TOF) Ratio to ≥0.8: Geometric Mean Analysis
Description: The efficacy analysis of TTR of participant TOF ratio to ≥0.8 was performed by estimating the geometric mean of TTR within each treatment group. TTR was monitored by applying electrical stimulations to the ulnar nerve every 15 seconds and assessing twitch response at the adductor pollicis muscle. T1 and T4 refer to magnitudes of the first and fourth twitches respectively, after nerve stimulation. The T4/T1 ratio (TOF; expressed as a decimal of up to 1.0) indicates the extent of recovery from NMB. A faster TTR of the TOF ratio to 0.8 indicates faster recovery from NMB. As specified by the protocol, analyses for this outcome measure were conducted in participants pooled by dosing method across depth of NMB (Sugammadex ABW [2 mg/kg ABW plus 4 mg/kg ABW] and Sugammadex IBW [2 mg/kg IBW plus 4 mg/kg IBW]) as well as in all randomized treatment arms separated by depth of NMB (Sugammadex 2 mg/kg ABW, Sugammadex 4 mg/kg ABW, Sugammadex 2 mg/kg IBW, and Sugammadex 4 mg/kg IBW).
Time Frame: Up to 69 minutes
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Sugammadex 2 mg/kg ABW | Sugammadex 4 mg/kg ABW | Sugammadex ABW (2 mg/kg ABW Plus 4 mg/kg ABW) | Sugammadex 2 mg/kg IBW | Sugammadex 4 mg/kg IBW | Sugammadex IBW (2 mg/kg IBW Plus 4 mg/kg IBW) | Neostigmine/Glycopyrrolate
Number analyzed (Participants) | 38 | 37 | 75 | 37 | 36 | 73 | 38
Minutes | 1.6 [1.3 to 1.8] | 1.5 [1.2 to 1.7] | 1.5 [1.3 to 1.7] | 2.5 [2.1 to 2.9] | 2.6 [2.1 to 3.1] | 2.5 [2.2 to 2.8] | 16.6 [12.8 to 21.7]
Statistical Analysis 1: Comparison: Sugammadex 2 mg/kg ABW vs Sugammadex 2 mg/kg IBW; Test type: Superiority; Ratio of geometric means = 0.63, 95% CI 2-sided [0.50 to 0.80] — Log transformation and t-distribution
Statistical Analysis 2: Comparison: Sugammadex 2 mg/kg ABW vs Neostigmine/Glycopyrrolate; Test type: Superiority; Ratio of geometric means = 0.09, 95% CI 2-sided [0.07 to 0.13] — Log transformation and t-distribution
Statistical Analysis 3: Comparison: Sugammadex 2 mg/kg IBW vs Neostigmine/Glycopyrrolate; Test type: Superiority; Ratio of geometric means = 0.15, 95% CI 2-sided [0.11 to 0.20] — Log transformation and t-distribution
Statistical Analysis 4: Comparison: Sugammadex 4 mg/kg ABW vs Sugammadex 4 mg/kg IBW; Test type: Superiority; Ratio of geometric means = 0.56, 95% CI 2-sided [0.44 to 0.72] — Log transformation and t-distribution
Statistical Analysis 5: Comparison: Sugammadex ABW (2 mg/kg ABW Plus 4 mg/kg ABW) vs Sugammadex IBW (2 mg/kg IBW Plus 4 mg/kg IBW); Test type: Superiority; Ratio of geometric means = 0.60, 95% CI 2-sided [0.51 to 0.70] — Log transformation and t-distribution

11. Secondary Outcome: Time to Recovery (TTR) of Participant Train of Four (TOF) Ratio to ≥0.7: Geometric Mean Analysis
Description: The efficacy analysis of TTR of participant TOF ratio to ≥0.7 was performed by estimating the geometric mean of TTR within each treatment group. TTR was monitored by applying electrical stimulations to the ulnar nerve every 15 seconds and assessing twitch response at the adductor pollicis muscle. T1 and T4 refer to magnitudes of the first and fourth twitches respectively, after nerve stimulation. The T4/T1 ratio (TOF; expressed as a decimal of up to 1.0) indicates the extent of recovery from NMB. A faster TTR of the TOF ratio to 0.7 indicates faster recovery from NMB. As specified by the protocol, analyses for this outcome measure were conducted in participants pooled by dosing method across depth of NMB (Sugammadex ABW [2 mg/kg ABW plus 4 mg/kg ABW] and Sugammadex IBW [2 mg/kg IBW plus 4 mg/kg IBW]) as well as in all randomized treatment arms separated by depth of NMB (Sugammadex 2 mg/kg ABW, Sugammadex 4 mg/kg ABW, Sugammadex 2 mg/kg IBW, and Sugammadex 4 mg/kg IBW).
Time Frame: Up to 61 minutes
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Sugammadex 2 mg/kg ABW | Sugammadex 4 mg/kg ABW | Sugammadex ABW (2 mg/kg ABW Plus 4 mg/kg ABW) | Sugammadex 2 mg/kg IBW | Sugammadex 4 mg/kg IBW | Sugammadex IBW (2 mg/kg IBW Plus 4 mg/kg IBW) | Neostigmine/Glycopyrrolate
Number analyzed (Participants) | 38 | 37 | 75 | 37 | 36 | 73 | 38
Minutes | 1.4 [1.2 to 1.6] | 1.3 [1.2 to 1.6] | 1.4 [1.2 to 1.5] | 2.1 [1.8 to 2.4] | 2.0 [1.7 to 2.5] | 2.1 [1.8 to 2.3] | 10.9 [8.1 to 14.6]
Statistical Analysis 1: Comparison: Sugammadex 2 mg/kg ABW vs Sugammadex 2 mg/kg IBW; Test type: Superiority; Ratio of geometric means = 0.66, 95% CI 2-sided [0.54 to 0.81] — Log transformation and t-distribution
Statistical Analysis 2: Comparison: Sugammadex 2 mg/kg ABW vs Neostigmine/Glycopyrrolate; Test type: Superiority; Ratio of geometric means = 0.13, 95% CI 2-sided [0.09 to 0.17] — Log transformation and t-distribution
Statistical Analysis 3: Comparison: Sugammadex 2 mg/kg IBW vs Neostigmine/Glycopyrrolate; Test type: Superiority; Ratio of geometric means = 0.19, 95% CI 2-sided [0.14 to 0.27] — Log transformation and t-distribution
Statistical Analysis 4: Comparison: Sugammadex 4 mg/kg ABW vs Sugammadex 4 mg/kg IBW; Test type: Superiority; Ratio of geometric means = 0.66, 95% CI 2-sided [0.52 to 0.83] — Log transformation and t-distribution
Statistical Analysis 5: Comparison: Sugammadex ABW (2 mg/kg ABW Plus 4 mg/kg ABW) vs Sugammadex IBW (2 mg/kg IBW Plus 4 mg/kg IBW); Test type: Superiority; Ratio of geometric means = 0.66, 95% CI 2-sided [0.57 to 0.77] — Log transformation and t-distribution

ADVERSE EVENTS:
Time Frame: Up to 14 days
Description: Analysis population consisted of all randomized participants who received at least one dose of study treatment.
Groups:
- Neostigmine + Glycopyrrolate: Following administration of NMBA, participants received a single i.v. bolus containing both Neostigmine (50 µg/kg; up to 5 mg maximum dose) and Glycopyrrolate (10 µg/kg; up to 1 mg maximum dose) as determined utilizing participant ABW. Neostigmine/Glycopyrrolate was used for reversal of moderate NMB. Active comparator treatment for reversal for deep NMB was not available.
Arm/Group | Sugammadex 2 mg/kg ABW | Sugammadex 4 mg/kg ABW | Sugammadex 2 mg/kg IBW | Sugammadex 4 mg/kg IBW | Neostigmine + Glycopyrrolate
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38 | 0/38 | 0/36 | 1/38
Serious Adverse Events (participants affected / at risk) | 1/38 | 0/38 | 3/38 | 4/36 | 3/38
Other Adverse Events (participants affected / at risk) | 36/38 | 32/38 | 36/38 | 32/36 | 32/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugammadex 2 mg/kg ABW (N=38) | Sugammadex 4 mg/kg ABW (N=38) | Sugammadex 2 mg/kg IBW (N=38) | Sugammadex 4 mg/kg IBW (N=36) | Neostigmine + Glycopyrrolate (N=38)
Cardiovascular insufficiency (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Borderline ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugammadex 2 mg/kg ABW (N=38) | Sugammadex 4 mg/kg ABW (N=38) | Sugammadex 2 mg/kg IBW (N=38) | Sugammadex 4 mg/kg IBW (N=36) | Neostigmine + Glycopyrrolate (N=38)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2) | 4 (4) | 3 (3) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4) | 1 (1) | 5 (5) | 4 (4) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (6) | 9 (10) | 10 (13) | 6 (6) | 7 (7)
Short-bowel syndrome (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 6 (6) | 1 (1) | 4 (4) | 2 (2) | 3 (3)
Neuromuscular block prolonged (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Procedural nausea (Injury, poisoning and procedural complications) | 9 (10) | 8 (8) | 4 (4) | 4 (4) | 5 (5)
Procedural pain (Injury, poisoning and procedural complications) | 28 (30) | 23 (23) | 28 (31) | 27 (27) | 24 (25)
Procedural vomiting (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 5 (5) | 1 (1) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 3 (3)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 3 (3) | 2 (2) | 2 (2) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (2):
  • Study Protocol (2018-07-05): https://cdn.clinicaltrials.gov/large-docs/70/NCT03346070/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/70/NCT03346070/SAP_001.pdf